CLINICAL TRIAL: NCT01253902
Title: Ocular Surface Tolerability Study of Prostaglandin Analogues in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMA-LUM-09-014
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Results first posted 2012-11-07 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-10

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost; Travoprost; Latanoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- bimatoprost ophthalmic solution 0.01% (Active Comparator): One drop of bimatoprost ophthalmic solution 0.01% (Lumigan®) administered to affected eye(s), once daily in the evening for 12 weeks.
  Interventions: Drug: bimatoprost ophthalmic solution 0.01%
- travoprost ophthalmic solution 0.004% (Active Comparator): One drop of travoprost ophthalmic solution 0.004% (Travatan Z®) administered to affected eye(s), once daily in the evening for 12 weeks.
  Interventions: Drug: travoprost ophthalmic solution 0.004%
- latanoprost ophthalmic solution 0.005% (Active Comparator): One drop of latanoprost ophthalmic solution 0.005% (Xalatan®) administered to affected eye(s), once daily in the evening for 12 weeks.
  Interventions: Drug: latanoprost ophthalmic solution 0.005%

INTERVENTIONS:
Drug: bimatoprost ophthalmic solution 0.01% — One drop of bimatoprost ophthalmic solution 0.01% administered to affected eye(s), once daily in the evening for 12 weeks.
  Other Names: Lumigan® 0.01%, Lumigan® RC
  Arms: bimatoprost ophthalmic solution 0.01%
Drug: travoprost ophthalmic solution 0.004% — One drop of travoprost ophthalmic solution 0.004% administered to affected eye(s), once daily in the evening for 12 weeks.
  Other Names: Travatan Z®
  Arms: travoprost ophthalmic solution 0.004%
Drug: latanoprost ophthalmic solution 0.005% — One drop of latanoprost ophthalmic solution 0.005% administered to affected eye(s), once daily in the evening for 12 weeks.
  Other Names: Xalatan®
  Arms: latanoprost ophthalmic solution 0.005%

SUMMARY:
This study evaluated the ocular surface tolerability of the prostaglandin analogues bimatoprost ophthalmic solution 0.01% (Lumigan® 0.01%), travoprost ophthalmic solution 0.004% (Travatan Z®) and latanoprost ophthalmic solution 0.005% (Xalatan®) in patients previously treated with Xalatan® who have open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ocular hypertension or open-angle glaucoma in at least 1 eye requiring treatment with an anti-glaucoma/ocular hypertensive medication
* Best corrected visual acuity score of 20/100 or better in both eyes
* Females on birth control pills must be on same type of pill and dose for at least 3 month

Exclusion Criteria:

* Use of Lumigan® 0.01%/Lumigan® RC, Lumigan®, Travatan® or Travatan Z® within 6 months
* History of or active ocular infection/inflammation (eg, uveitis)
* Punctal plug use
* Required use of ocular medications during the study other than study medication (intermittent use of certain types artificial tears acceptable)
* Intraocular surgery or glaucoma laser surgery in study eye(s) within 3 months
* History of corneal refractive laser surgery (eg, LASIK, LASEK) in study eye(s)
* Planned contact lens wear during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Rogers, Arkansas, United States
- Calgary, Alberta, Canada

REFERENCES:
- [Derived] Schwartz GF, Hollander DA, Williams JM. Evaluation of eye drop administration technique in patients with glaucoma or ocular hypertension. Curr Med Res Opin. 2013 Nov;29(11):1515-22. doi: 10.1185/03007995.2013.833898. Epub 2013 Sep 5. PMID 24006861
- [Derived] Crichton AC, Vold S, Williams JM, Hollander DA. Ocular surface tolerability of prostaglandin analogs and prostamides in patients with glaucoma or ocular hypertension. Adv Ther. 2013 Mar;30(3):260-70. doi: 10.1007/s12325-013-0014-7. Epub 2013 Mar 7. PMID 23475405

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost Ophthalmic Solution 0.01% | Travoprost Ophthalmic Solution 0.004% | Latanoprost Ophthalmic Solution 0.005%
Started | 56 | 53 | 55
Completed | 51 | 51 | 51
Not Completed | 5 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost Ophthalmic Solution 0.01% | Travoprost Ophthalmic Solution 0.004% | Latanoprost Ophthalmic Solution 0.005% | Total
Number analyzed (Participants) | 56 | 53 | 55 | 164
Age Continuous [Mean (Standard Deviation); unit: Years] | 65.1 (11.76) | 63.2 (13.57) | 64.7 (12.28) | 64.3 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 25 | 31 | 92
  Male | 20 | 28 | 24 | 72

OUTCOME MEASURES:

1. Primary Outcome: Mean Conjunctival Hyperemia at Week 12
Description: Conjunctival hyperemia was analyzed using the average of the scores of both eyes. Hyperemia is engorgement of the blood vessels (redness) of the bulbar conjunctiva of the eye (the clear membrane covering the white surface of the eye). Hyperemia was graded on a 5 point scale where 0=none (normal), 0.5=trace (trace flush reddish pink), 1=Mild (mild flush reddish color), 2=Moderate (bright red color) and 3=severe (deep bright diffuse redness).
Time Frame: Week 12
Population: Intent-to-treat population (ITT) included all participants who were randomized to study medication.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Bimatoprost Ophthalmic Solution 0.01% | Travoprost Ophthalmic Solution 0.004% | Latanoprost Ophthalmic Solution 0.005%
Number analyzed (Participants) | 56 | 53 | 55
Score on a scale | 0.42 (0.48) | 0.46 (0.44) | 0.44 (0.57)

2. Secondary Outcome: Mean Corneal Staining With Fluorescein at Week 12
Description: Corneal staining was analyzed using the average of the scores of both eyes. The cornea is the transparent front part of the eye which covers the iris and pupil. To detect the presence or absence of corneal puncta (tiny disruptions in the surface of the eye), fluorescein dye is administered into the eye and the eye is graded using a 5-point scale where 0=None (no puncta), 0.5=Trace (1-5 puncta), 1=Mild (6-20 puncta), 2=Moderate (>20 puncta) and 3=Severe (too many puncta to count).
Time Frame: Week 12
Population: Intent-to-treat (ITT) population included all participants who were randomized and received study medication.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Bimatoprost Ophthalmic Solution 0.01% | Travoprost Ophthalmic Solution 0.004% | Latanoprost Ophthalmic Solution 0.005%
Number analyzed (Participants) | 56 | 53 | 55
Score on a scale | 0.31 (0.45) | 0.32 (0.48) | 0.22 (0.30)

3. Secondary Outcome: Mean Tear Break Up Time (TBUT) at Week 12
Description: Tear Break Up Time was analyzed using the average of the readings of both eyes. TBUT is defined as the time (seconds) required for dry spots to appear on the surface of the eye after blinking. The longer it takes, the more stable the tear film.
Time Frame: Week 12
Population: Intent-to-treat (ITT) population included all participants who were randomized and received study medication.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Bimatoprost Ophthalmic Solution 0.01% | Travoprost Ophthalmic Solution 0.004% | Latanoprost Ophthalmic Solution 0.005%
Number analyzed (Participants) | 56 | 53 | 55
Seconds | 9.7 (5.71) | 9.7 (4.96) | 9.3 (4.04)

ADVERSE EVENTS:
Arm/Group | Bimatoprost Ophthalmic Solution 0.01% | Travoprost Ophthalmic Solution 0.004% | Latanoprost Ophthalmic Solution 0.005%
Serious Adverse Events (participants affected / at risk) | 1/56 | 1/53 | 3/55
Other Adverse Events (participants affected / at risk) | 0/56 | 0/53 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Ophthalmic Solution 0.01% (N=56) | Travoprost Ophthalmic Solution 0.004% (N=53) | Latanoprost Ophthalmic Solution 0.005% (N=55)
Gastrointestinal Bleed (Gastrointestinal disorders) | 0 | 0 | 1
Aspiration Pneumonia resulting in death (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Punctured colon (Gastrointestinal disorders) | 0 | 0 | 1
Infection from Punctured colon (Infections and infestations) | 0 | 0 | 1
Branch retinal artery occlusion (Eye disorders) | 1 | 0 | 0
Transient Ischemic Attack (Vascular disorders) | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.